CLINICAL TRIAL: NCT04693234
Title: Phase 2 Study Investigating Efficacy and Safety of Anti-PD-1 Monoclonal Antibody Tislelizumab (BGB-A317) Combined With or Without Anti-TIGIT Monoclonal Antibody BGB-A1217 in Patients With Previously Treated Recurrent or Metastatic Cervical Cancer
Brief Title: AdvanTIG-202: Anti-PD-1 Monoclonal Antibody Tislelizumab (BGB-A317) Combined With or Without Anti-TIGIT Monoclonal Antibody Ociperlimab (BGB-A1217) in Participants With Previously Treated Recurrent or Metastatic Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-A1217-202; 2020-004657-77 (EudraCT Number); AdvanTIG-202 (Other: BeiGene); CTR20212809 (Other: ChinaDrugTrials); CTR20210588 (Other: ChinaDrugTrials)
Record Dates: First submitted 2020-12-22; First posted 2021-01-05 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: Ociperlimab + Tislelizumab (Experimental): Tislelizumab 200 milligrams (mg) intravenously (IV) once every 3 weeks (Q3W) combined with ociperlimab (BGB-A1217) 900 mg IV Q3W
  Interventions: Biological: Tislelizumab; Biological: Ociperlimab
- Cohort 2: Tislelizumab (Experimental): Tislelizumab 200 mg IV Q3W monotherapy
  Interventions: Biological: Tislelizumab

INTERVENTIONS:
Biological: Tislelizumab — 200 mg administered intravenously once every 3 weeks on day 1 of each cycle
  Other Names: BGB-A317; TEVIMBRA®
Biological: Ociperlimab — 900 mg administered intravenously once every 3 weeks on day 1 of each cycle
  Other Names: BGB-A1217
  Arms: Cohort 1: Ociperlimab + Tislelizumab

SUMMARY:
This study tested how well and how safely the drug tislelizumab, given either alone or with another drug called ociperlimab (BGB-A1217), worked in people with cervical cancer that had come back or spread after previous treatments. The study included two groups and took place at multiple medical centers.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix.
2. Progression on or after one or more lines of chemotherapy for management of recurrent or metastatic disease and is not amenable to curative treatment (eg, systemic chemotherapy, surgery, or radiotherapy).
3. Measurable disease as assessed by RECIST v1.1. Note: A lesion in an area subjected to prior loco-regional therapy, including previous radiotherapy, is not considered measurable unless there has been demonstrated progression in the lesion since the therapy as defined by RECIST v1.1.
4. Participants must submit qualified archival tumor tissue (formalin-fixed paraffin-embedded block containing tumor [preferred] or approximately 15 [at least 6] unstained slides) with an associated pathology report, or agree to a tumor biopsy for determination of Programmed death-ligand 1 (PD-L1) expression and other biomarker analyses (fresh tumor biopsies are strongly recommended at baseline in participants with readily accessible tumor lesions and who consent to the biopsies).
5. Participant must have adequate organ function as indicated by the screening laboratory values obtained within 7 days before the first study treatment.

Exclusion Criteria:

1. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, TIGIT or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways.
2. Any active malignancy ≤ 2 years before first dose of study drug except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of breast).
3. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage (recurrence within 2 weeks of intervention).
4. Any major surgical procedure ≤ 28 days before first dose of study drug. Participants must have recovered adequately from the toxicity and/or complications from the intervention before the first dose of study drug.
5. Has received any chemotherapy, immunotherapy (eg, interleukin, interferon, thymosin, etc.) or any investigational therapies within 14 days or 5 half-lives (whichever is longer) before the first dose of study drug or has received palliative radiation treatment or other local regional therapies within 14 days before the first dose of study drug.

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 178 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (68):
- Bulgaria (4):
  - "Mhat uni hospital" ood, Panagyurishte
  - Complex Oncology Center Rousse Eood, Rousse
  - Medical center nadezhda clinical eood, Sofia
  - Acibadem city clinic tokuda umhat ead, department of medical oncology, Sofia
- China (28):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Sun yat-sen memorial hospital, sun yat-sen university (south), Guanzhou, Guangdong
  - The Tumor Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - Hainan Cancer Hospital, Haikou, Hainan
  - Henan Cancer Hospital - Oncology, Zhengzhou, Henan
  - Hubei Cancer Hospital - Oncology, Wuhan, Hubei
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital - GCP Office, Changsha, Hunan
  - Xuzhou Cancer Hospital, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Jilin Guowen Hospital, Jilin, Jilin
  - Liaoning Cancer Hospital & Institute - Medical Oncology - Oncology, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Second Hospital Of Shanxi Medical University, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Tianjin Medical University Cancer institute & Hospital, Tianjin, Tianjin Municipality
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Beijing Cancer Hosptial, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Linyi Cancer Hospital, Shandong
  - The First Affiliated Hospital of Xiamen University - Oncology, Xiamen
- Poland (2):
  - Szpitale Pomorskie Spółka z ograniczoną odpowiedzialnością, Gdynia
  - Przychodnia lekarska komed, Konin
- Russia (6):
  - State healthcare institution oncologic dispensary no. 2 - health department of krasnodar region, Krasnodar, Krasnodarskiy Kray
  - Fsbi of higher education"ogarev mordovia state university", Saransk, Mordovia Republic
  - Oncological Scientific Center LLC, Pesochny, Sankt-Peterburg
  - Sbhi of stavropol region "pyatigorsk interdistrict oncologic dispensary", Pyatigorsk, Stavropol Kray
  - Arkhangelsk regional clinical oncological dispensary, Arkhangelsk
  - State budgetary healthcare institution-chelyabinsk regional clinical center of oncology and nuclear, Chelyabinsk
- South Korea (12):
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyemyung University Dongsan Hospital, Daegu
  - Ajou University Hospital, Gyeonggi-do
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea Institute of Radiological & Medical Sciences, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Taiwan (6):
  - Chi Mei Hospital, Liouying, Tainan
  - Linkou Chang Gung Memorial Hospital, Tainan
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (4):
  - Siriraj Hospital, Bangkok Noi, Bangkok
  - Songklanagarind Hospital, Prince of Songkla University, Hat Yai
  - Srinagarind Hospital (Khon Kaen University), Khon Kaen
  - Phramongkutklao Hospital, Ratchathewi
- Ukraine (6):
  - Public Non-Profit Institution "Precarpathian Oncology Center Of Ivano-Frankivsk Regional Council", Ivano-Frankivsk Oblast, Ivano-Frankivsk Oblast
  - Medical and diagnostic center of private enterprise private production company "acinus", Kirovograd, Kirovohrad Oblast
  - Communal Non-Profit Enterprise Of Sumy Regional Council Sumy Regional Clinical Oncological Dispensar, Sumy, Sumska Oblast
  - National Cancer Institute, Kiev
  - Medical center of llc oncolife, Kropyvnytskyi
  - Volyn Regional Medical Center Of Oncology, Lutsk

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Lee JY, Boonyapipat S, Yuan G, Kim HS, Lee JW, Wang L, Wang T, Wang D, Yao D, Liu H, Chang CL, Andabekov TT, Zhang X, Wang W, Kim YM, Sinielnikov IV, Wang K, Gao Y, Mu X, Wu L. AdvanTIG-202: Phase 2 open-label, two-cohort multicenter study of ociperlimab plus tislelizumab and tislelizumab alone in patients with previously treated recurrent or metastatic cervical cancer. Gynecol Oncol. 2025 Jul;198:25-32. doi: 10.1016/j.ygyno.2025.04.579. Epub 2025 May 23. PMID 40411966

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in multiple study centers in China, South Korea, and Europe.The first participant dosed was on March 3rd, 2021 and the last participant completed on August 31st, 2023.
Pre-assignment Details: The study was composed of an initial screening phase (up to 28 days), a treatment phase, an end of treatment visit, an on-site Safety Follow-up Visit, and 2 Safety Follow-up Visits by telephone after the last dose of study treatment.
Groups:
- Cohort 1: Ociperlimab + Tislelizumab: Participants received tislelizumab 200 milligrams (mg) intravenously (IV) and ociperlimab 900 mg IV once every 3 weeks (Q3W) until disease progression, unacceptable toxicity, or withdrawal of consent.
- Cohort 2: Tislelizumab: Participants received tislelizumab 200 mg administered intravenously once every 3 weeks until disease progression, unacceptable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab | Cohort 2: Tislelizumab
Started | 138 | 40
Completed | 0 | 0
Not Completed | 138 | 40
Not completed — Death | 79 | 19
Not completed — Sponsor Ended Study | 47 | 18
Not completed — Withdrawal by Subject | 10 | 2
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set is defined as all participants who received >= 1 dose of any study drug for each cohort.
Groups:
- Cohort 1: Ociperlimab + Tislelizumab: Participants received tislelizumab 200 mg IV and ociperlimab 900 mg IV once every 3 weeks until disease progression, unacceptable toxicity, or withdrawal of consent.
- Cohort 2: Tislelizumab: Participants received tislelizumab 200 mg IV once every 3 weeks until disease progression, unacceptable toxicity, or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab | Cohort 2: Tislelizumab | Total
Number analyzed (Participants) | 138 | 40 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (10.28) | 51.2 (9.74) | 52.3 (10.15)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 138 | 40 | 178
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 117 | 37 | 154
  White | 21 | 3 | 24
Region of Enrollment [Number; unit: participants]
  China | 71 | 17 | 88
  South Korea | 30 | 8 | 38
  Taiwan | 10 | 6 | 16
  Ukraine | 10 | 0 | 10
  Russia | 8 | 3 | 11
  Thailand | 6 | 6 | 12
  Bulgaria | 2 | 0 | 2
  Poland | 1 | 0 | 1
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — The ECOG scale assesses disease status from 0 to 5. A score of 0 means fully active with no restrictions, while 1 indicates limitations in strenuous activities but the ability to do light work. Score 2 signifies ambulatory and capable of self-care, yet unable to work, being active for over 50% of waking hours. Score 3 reflects limited self-care, confined to bed or a chair for more than half the day. Score 4 indicates complete disability, with the participant fully bedbound, and score 5 means deceased.
  Participants
    0 | 53 | 16 | 69
    1 | 85 | 24 | 109
Programmed Death-Ligand 1 (PD-L1) Expression [Count of Participants; unit: Participants] — PD-L1 is a protein found in higher-than-normal amounts on some types of cancer cells which can prevent the body's immune cells from killing the PD-L1-containing cancer cells.
  PD-L1 score was defined by the total percentage of the tumor area (tumor and any desmoplastic stroma) covered by tumor cells and tumor-associated immune cells with PD-L1 staining at any intensity as visually estimated based on Tumor Area Positive [TAP] Score methodology. (TAP score methodology had been previously referred to as the visually-estimated Combined Positive Score [vCPS] score).
  Participants
    PD-L1 Score >= 5% | 84 | 20 | 104
    PD-L1 Score < 5% | 53 | 20 | 73
    Not Evaluable | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Objective Response Rate (ORR) Assessed by an Independent Review Committee (IRC) in PD-L1-Positive Participants
Description: ORR is defined as the percentage of participants who had confirmed complete response (CR) or partial response (PR) as assessed by the IRC per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1).
  PD-L1-positive refers to participants whose tumors had a PD-L1 TAP score ≥ 5%.
Time Frame: Up to the primary efficacy analysis data cut-off date on June 16, 2022, the median follow-up duration was 7.36 months for Cohort 1.
Population: The PD-L1 Score ≥ 5% Safety Analysis Set includes all treated participants whose tumors had PD-L1 TAP Score ≥ 5%.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab
Number analyzed (Participants) | 84
percentage of participants | 26.2 [17.2 to 36.9]
Statistical Analysis 1: Comparison: Cohort 1: Ociperlimab + Tislelizumab; Test type: Superiority; p = 0.0054, Binomial Exact Test; The p-value was calculated from the binomial exact test of tislelizumab combined with ociperlimab versus historical rate of 0.15

2. Primary Outcome: Cohort 1: ORR Assessed by the IRC in All Treated Participants
Description: ORR is defined as the percentage of participants who had a confirmed CR or PR as assessed by the IRC per RECIST v1.1.
Time Frame: as for outcome 1
Population: The Safety Analysis Set includes all participants who received at least 1 dose of any study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab
Number analyzed (Participants) | 138
percentage of participants | 22.5 [15.8 to 30.3]
Statistical Analysis 1: Comparison: Cohort 1: Ociperlimab + Tislelizumab; Test type: Superiority; p = 0.0127, Binomial Exact Test; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Cohort 2: Objective Response Rate (ORR) Assessed by an Independent Review Committee in All Treated Participants
Description: ORR is defined as the percentage of participants who had confirmed complete response (CR) or partial response (PR) as assessed by the IRC per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1).
Time Frame: Up to the primary efficacy analysis data cut-off date on June 16, 2022, the median follow-up duration was 10.40 months for Cohort 2.
Population: The Safety Analysis Set includes all participants who received at least 1 dose of any study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: Tislelizumab
Number analyzed (Participants) | 40
percentage of participants | 32.5 [18.6 to 49.1]

4. Secondary Outcome: ORR Assessed by the Investigator in PD-L1-Positive Participants
Description: ORR is defined as the percentage of participants who had confirmed CR or PR as assessed by the investigator per RECIST v1.1 in the PD-L1 Score >= 5% Safety Analysis Set.
Time Frame: Up to the primary efficacy analysis data cut-off date on June 16, 2022, the median follow-up duration was 7.36 months for Cohort 1 and 10.40 months for Cohort 2.
Population: The PD-L1 Score ≥ 5% Safety Analysis Set includes all treated participants whose tumors had PD-L1 Score ≥ 5%.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab | Cohort 2: Tislelizumab
Number analyzed (Participants) | 84 | 20
percentage of participants | 25.0 [16.2 to 35.6] | 30 [11.9 to 54.3]

5. Secondary Outcome: ORR as Assessed by the Investigator in All Treated Participants
Description: ORR is defined as the percentage of participants who had a confirmed CR or PR as assessed by the investigator per RECIST v1.1.
Time Frame: as for outcome 4
Population: The Safety Analysis Set includes participants who received at least 1 dose of any study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab | Cohort 2: Tislelizumab
Number analyzed (Participants) | 138 | 40
percentage of participants | 21.0 [14.5 to 28.8] | 22.5 [10.8 to 38.5]

6. Secondary Outcome: Duration of Response (DOR) Assessed by the IRC
Description: DOR is defined as the time from the first confirmed objective response until the first documentation of progression or death, whichever occurred first, assessed by the IRC according to RECIST v1.1 in the Safety Analysis Set.
Time Frame: as for outcome 4
Population: Safety Analysis Set. Only participants with best overall response of complete response or partial response confirmed per RECIST v1.1 by the IRC were included in the analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab | Cohort 2: Tislelizumab
Number analyzed (Participants) | 31 | 13
Months | NA [5.6 to NA] — Not estimable due to insufficient number of participants with events | NA [4.1 to NA] — Not estimable due to insufficient number of participants with events

7. Secondary Outcome: Duration of Response (DOR) Assessed by the Investigator
Description: DOR is defined as the time from the first confirmed objective response until the first documentation of progression or death, whichever comes first, assessed by the investigator according to RECIST v1.1 in the Safety Analysis Set. Data was based on number of responders.
Time Frame: as for outcome 4
Population: Safety Analysis Set. Only participants with best overall response of complete response or partial response confirmed per RECIST v1.1 by the investigator were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab | Cohort 2: Tislelizumab
Number analyzed (Participants) | 29 | 9
Months | NA [5.5 to NA] — Not estimable due to insufficient number of participants with events | NA [5.6 to NA] — Not estimable due to insufficient number of participants with events

8. Secondary Outcome: Progression Free Survival (PFS)
Description: Defined as the time from the date of first dose of study drug to the date of first documentation of disease progression or death, whichever occurred first as assessed by both the IRC and the investigator's review per RECIST v1.1 in the Safety Analysis Set.
Time Frame: as for outcome 4
Population: Safety Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab | Cohort 2: Tislelizumab
Number analyzed (Participants) | 138 | 40
Months
  IRC | 3.5 [2.6 to 4.9] | 5.7 [2.3 to 8.1]
  Investigator | 3.9 [2.6 to 4.4] | 5.7 [2.6 to 9.2]

9. Secondary Outcome: Time to Response (TTR) Assessed by the IRC
Description: TTR is defined as the time from the date of first dose of study drug to the first documentation of response as assessed by the IRC per RECIST v1.1, in the Safety Analysis Set.
Time Frame: Up to the primary efficacy analysis data cut-off date on June 16, 2022, the median follow-up was 7.36 months for Cohort 1 and 10.40 months for Cohort 2.
Population: The Safety Analysis Set. Only participants with best overall response of complete response or partial response confirmed by the IRC per RECIST v1.1 were included in the analysis.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab | Cohort 2: Tislelizumab
Number analyzed (Participants) | 31 | 13
Weeks | 9.02 (4.704) | 11.78 (4.709)

10. Secondary Outcome: Time to Response (TTR) Assessed by the Investigator
Description: TTR is defined as the time from the date of first dose of study drug to the first documentation of response as assessed by the investigator per RECIST v1.1, in the Safety Analysis Set.
Time Frame: as for outcome 9
Population: The Safety Analysis Set. Only participants with best overall response of complete response or partial response confirmed by the investigator per RECIST v1.1 were included in the analysis.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab | Cohort 2: Tislelizumab
Number analyzed (Participants) | 29 | 9
Weeks | 10.66 (3.010) | 8.92 (3.174)

11. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants who achieve CR, PR, or stable disease (SD) as assessed by both the IRC and investigator per RECIST v1.1 in the Safety Analysis Set.
Time Frame: as for outcome 4
Population: The Safety Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab | Cohort 2: Tislelizumab
Number analyzed (Participants) | 138 | 40
percentage of participants
  IRC | 63.0 [54.4 to 71.1] | 67.5 [50.9 to 81.4]
  Investigator | 62.3 [53.7 to 70.4] | 75.0 [58.8 to 87.3]

12. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Defined as the percentage of participants who achieve CR, PR, or durable SD (SD ≥ 24 weeks) as assessed by both the IRC and investigator per RECIST v1.1 in the Safety Analysis Set.
Time Frame: as for outcome 4
Population: The Safety Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 2: Tislelizumab: Participants received tislelizumab 200 mg IV and ociperlimab 900 mg IV once every 3 weeks until disease progression, unacceptable toxicity, or withdrawal of consent.
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab | Cohort 2: Tislelizumab
Number analyzed (Participants) | 138 | 40
percentage of participants
  IRC | 29.0 [21.6 to 37.3] | 50.0 [33.8 to 66.2]
  Investigator | 31.2 [23.6 to 39.6] | 50.0 [33.8 to 66.2]

13. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of randomization to the date of death due to any cause. Median OS was estimated using Kaplan-Meier methodology.
Time Frame: as for outcome 4
Population: The Safety Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab | Cohort 2: Tislelizumab
Number analyzed (Participants) | 138 | 40
Months | 9.0 [8.1 to 10.4] | NA [10.5 to NA] — Not estimable due to insufficient number of participants with events

14. Secondary Outcome: Mean Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status/Quality of Life, Physical Functioning, and Pain Scores
Description: The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 = Not at all (best) and 4 = Very Much (worst) and 2 global health quality of life (QOL) questions answered on a 7-point scale where 1 = Very poor and 7 = Excellent. Raw scores are transformed into a 0 to 100 scale via linear transformation. Higher scores in GHS and functional scales indicate better quality of life. Lower scores in symptom scales indicate better quality of life.
Time Frame: Baseline to Cycles 3 and 5 ( Each cycle was 21 days)
Population: The Safety Analysis Set with available EORTC QLQ-C30 values at Baseline; Only participants with data at baseline and at each time point are included.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab | Cohort 2: Tislelizumab
Number analyzed (Participants) | 122 | 38
Score on a scale
  GHS/QoL: Baseline Score | 64.21 (20.821) | 62.06 (22.402)
  GHS/QoL: Change from Baseline to Cycle 3 Day 1: number analyzed (Participants) | 112 | 33
  GHS/QoL: Change from Baseline to Cycle 3 Day 1 | 0.37 (22.158) | 5.30 (23.088)
  GHS/QoL: Change from Baseline to Cycle 5 Day 1: number analyzed (Participants) | 77 | 26
  GHS/QoL: Change from Baseline to Cycle 5 Day 1 | 3.46 (18.355) | 5.13 (21.995)
  Physical Functioning: Baseline Score | 78.91 (19.211) | 76.67 (22.501)
  Physical Functioning: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 112 | 33
  Physical Functioning: Change from Baseline at Cycle 3 Day 1 | -2.62 (16.582) | 1.82 (18.876)
  Physical Functioning: Change from Baseline at Cycle 5 Day 1: number analyzed (Participants) | 76 | 26
  Physical Functioning: Change from Baseline at Cycle 5 Day 1 | 0.00 (14.927) | 5.38 (16.113)
  Pain: Baseline Score | 27.73 (28.070) | 30.26 (27.084)
  Pain: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 112 | 33
  Pain: Change from Baseline at Cycle 3 Day 1 | -2.08 (21.820) | -9.09 (26.051)
  Pain: Change from Baseline at Cycle 5 Day 1: number analyzed (Participants) | 77 | 26
  Pain: Change from Baseline at Cycle 5 Day 1 | -2.16 (22.353) | -8.97 (24.599)

15. Secondary Outcome: Mean Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Symptom Specific Scale for Cervical Cancer (EORTC QLQ-CX24) Index Score
Description: QLQ-CX24 is the cervical cancer module of the QLQ-C30. CX24 is comprised of 24 questions grouped into 3 symptom scales and 6 single symptom items. Each question is answered on a scale from 1 (not at all) to 4 (very much). The scales include Symptom Experience (11 items), Body Image (3 items) and Sexual/vaginal Functioning (4 items). The single symptom items include Lymphedema, Peripheral Neuropathy, Menopausal Symptoms, Sexual Worry, Sexual Activity and Sexual Enjoyment. Raw scores are transformed into a 0 to 100 scale via linear transformation. The Index score is calculated as the average of the 3 symptom scales and 6 single item scores. Lower scores indicate better HRQoL.
Time Frame: Baseline to Cycles 3 and 5 ( Each cycle was 21 days)
Population: The Safety Analysis Set with available EORTC QLQ-CX24 values at Baseline; Only participants with data at baseline and at each time point are included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab | Cohort 2: Tislelizumab
Number analyzed (Participants) | 122 | 38
score on a scale
  Baseline Score | 30.86 (6.942) | 31.43 (4.497)
  Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 112 | 33
  Change from Baseline at Cycle 3 Day 1 | 0.61 (5.915) | -0.71 (4.163)
  Change from Baseline at Cycle 5 Day 1: number analyzed (Participants) | 77 | 26
  Change from Baseline at Cycle 5 Day 1 | -0.15 (5.790) | 1.05 (4.227)

16. Secondary Outcome: Number of Participants Experiencing Treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drugs, whether considered related to study drugs or not.
  An SAE is any untoward medical occurrence that, at any dose:
  * Resulted in death
  * Was life-threatening
  * Required hospitalization or prolongation of existing hospitalization
  * Resulted in disability/incapacity
  * Was a congenital anomaly/birth defect
  * Was considered a significant medical AE by the investigator based on medical judgement (eg, may jeopardize the patient or may require medical/surgical intervention to prevent one of the outcomes listed above).
Time Frame: From the first dose of study drug to 30 days after the last dose; maximum treatment exposure was 23.5 months.
Population: The Safety Analysis Set includes all participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab | Cohort 2: Tislelizumab
Number analyzed (Participants) | 138 | 40
Participants
  Number of Participants with at least one TEAE | 135 | 39
  Number of participants with at least one SAE | 61 | 17

17. Secondary Outcome: Serum Ociperlimab (BGB-A1217) Concentrations at Specified Timepoints
Description: The timepoints are defined as predose (within 60 minutes before starting infusion) and postdose (within 30 minutes after the end of infusion).
Time Frame: Day 1 of Cycles 1, 2, 5, 9, and 17 (each cycle was 21 days)
Population: The Pharmacokinetic Analysis (PK) Set includes all participants who received at least 1 dose of any component of study drug per the protocol, for whom any post-dose PK data are available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Cohort 1 (Predose): Ociperlimab: 900 mg administered intravenously once every 3 weeks on day 1 of each cycle. Predose was collected within 60 minutes before starting infusion
- Cohort 1 (Postdose): Ociperlimab: 900 mg administered intravenously once every 3 weeks on day 1 of each cycle. Postdose was collected within 30 minutes after the end of infusion.
Arm/Group | Cohort 1 (Predose) | Cohort 1 (Postdose)
Number analyzed (Participants) | 138 | 138
μg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 138 | 134
  Cycle 1 Day 1 | 0.00 (NA) — Not estimable since all values were below the limit of quantitation | 363.19 (24.21)
  Cycle 2 Day 1: number analyzed (Participants) | 119 | 0
  Cycle 2 Day 1 | 46.60 (46.98) |
  Cycle 5 Day 1: number analyzed (Participants) | 67 | 71
  Cycle 5 Day 1 | 82.57 (55.30) | 440.70 (25.35)
  Cycle 9 Day 1: number analyzed (Participants) | 41 | 0
  Cycle 9 Day 1 | 89.13 (56.58) |
  Cycle 17 Day 1: number analyzed (Participants) | 24 | 0
  Cycle 17 Day 1 | 88.84 (63.62) |

18. Secondary Outcome: Serum Tislelizumab Concentrations at Specified Timepoints
Description: as for outcome 17
Time Frame: Day 1 of Cycles 1, 2, 5, 9, and 17 (each cycle is 21 days)
Population: The Pharmacokinetic Analysis Set includes all participants who received >= 1 dose of any component of study drug per the protocol, for whom any post-dose PK data are available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Cohort 1 (Predose); Cohort 2 (Predose): Tislelizumab: 200 mg administered intravenously once every 3 weeks on day 1 of each cycle. Predose was collected within 60 minutes before starting infusion
- Cohort 1 (Postdose); Cohort 2 (Postdose): Tislelizumab: 200 mg administered intravenously once every 3 weeks on day 1 of each cycle. Postdose was collected within 30 minutes after the end of infusion.
Arm/Group | Cohort 1 (Predose) | Cohort 1 (Postdose) | Cohort 2 (Predose) | Cohort 2 (Postdose)
Number analyzed (Participants) | 138 | 138 | 40 | 40
μg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 136 | 136 | 40 | 40
  Cycle 1 Day 1 | 0.00 (NA) — Not estimable since all values were below the limit of quantitation | 77.38 (21.78) | 0.00 (NA) — Not estimable since all values were below the limit of quantitation | 84.24 (18.19)
  Cycle 2 Day 1: number analyzed (Participants) | 121 | 0 | 37 | 0
  Cycle 2 Day 1 | 17.86 (35.69) |  | 20.03 (36.62) |
  Cycle 5 Day 1: number analyzed (Participants) | 68 | 73 | 24 | 24
  Cycle 5 Day 1 | 36.66 (44.97) | 113.80 (24.68) | 41.51 (42.89) | 128.48 (24.06)
  Cycle 9 Day 1: number analyzed (Participants) | 41 | 0 | 21 | 0
  Cycle 9 Day 1 | 42.84 (46.50) |  | 56.78 (28.55) |
  Cycle 17 Day 1: number analyzed (Participants) | 27 | 0 | 12 | 0
  Cycle 17 Day 1 | 45.16 (55.71) |  | 56.25 (21.56) |

19. Secondary Outcome: Number of Participants Who Developed Positive Anti-drug Antibodies (ADAs) to Ociperlimab
Description: Number and percentage of participants who developed detectable ADAs to ociperlimab during the treatment period.
Time Frame: Samples for ADA analysis were collected predose on Day 1 of Cycles 1, 2, 5, 9 and 17, and at the Safety Follow-up Visit (30 days after last dose) up to the immunogenicity data cut-off date of June 1, 2023 (approximately 21 months).
Population: The ADA Analysis Set includes all participants who received at least 1 dose of any component of study drug for whom both baseline antidrug antibody result and at least 1 post-baseline antidrug antibody result were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab
Number analyzed (Participants) | 127
Participants | 0

20. Secondary Outcome: Number of Participants Who Developed Anti-drug Antibodies (ADAs) to Tislelizumab
Description: Number and percentage of participants who developed detectable ADAs during the treatment period.
Time Frame: Samples for ADA analysis were collected predose on Day 1 of Cycles 1, 2, 5, 9 and 17, and at the Safety Follow-up Visit (30 days after last dose), up to the immunogenicity data cut-off date of June 1, 2023 (approximately 21 months).
Population: The ADA Analysis Set includes all participants who received at least 1 dose of any component of study drug for whom both baseline antidrug antibody result and at least 1 post-baseline antidrug antibody result are available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab | Cohort 2: Tislelizumab
Number analyzed (Participants) | 127 | 39
Participants | 19 | 7

ADVERSE EVENTS:
Time Frame: All-cause mortality: From randomization through the end of study; up to 24.5 months. Adverse events: From the first dose to 30 days after the last dose; maximum treatment exposure was 23.5 months.
Arm/Group | Cohort 1: Ociperlimab + Tislelizumab | Cohort 2: Tislelizumab
All-Cause Mortality (participants affected / at risk) | 79/138 | 19/40
Serious Adverse Events (participants affected / at risk) | 61/138 | 17/40
Other Adverse Events (participants affected / at risk) | 128/138 | 37/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Ociperlimab + Tislelizumab (N=138) | Cohort 2: Tislelizumab (N=40)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 3 (5) | 2 (2)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 4 (4) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (6) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 3 (3)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Retroperitoneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 11 (12) | 2 (5)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 4 (5) | 3 (3)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urogenital fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Ociperlimab + Tislelizumab (N=138) | Cohort 2: Tislelizumab (N=40)
Anaemia (Blood and lymphatic system disorders) | 48 (66) | 15 (23)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 4 (4) | 3 (3)
Hypothyroidism (Endocrine disorders) | 27 (28) | 8 (9)
Abdominal pain (Gastrointestinal disorders) | 9 (11) | 6 (7)
Abdominal pain lower (Gastrointestinal disorders) | 9 (15) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 9 (9) | 1 (1)
Constipation (Gastrointestinal disorders) | 18 (20) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 15 (18) | 2 (4)
Dyspepsia (Gastrointestinal disorders) | 5 (6) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 27 (34) | 6 (7)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 17 (22) | 3 (3)
Asthenia (General disorders) | 8 (12) | 3 (6)
Chills (General disorders) | 11 (11) | 1 (1)
Fatigue (General disorders) | 8 (10) | 2 (2)
Influenza like illness (General disorders) | 2 (2) | 3 (3)
Malaise (General disorders) | 6 (6) | 1 (2)
Oedema peripheral (General disorders) | 6 (7) | 1 (1)
Pyrexia (General disorders) | 27 (38) | 7 (7)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 2 (3)
COVID-19 (Infections and infestations) | 10 (11) | 3 (3)
Urinary tract infection (Infections and infestations) | 16 (18) | 10 (11)
Alanine aminotransferase increased (Investigations) | 16 (24) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 24 (35) | 5 (6)
Blood alkaline phosphatase increased (Investigations) | 12 (14) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 3 (3)
Blood creatinine increased (Investigations) | 16 (25) | 6 (6)
Blood lactate dehydrogenase increased (Investigations) | 2 (4) | 4 (4)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 5 (5)
Blood thyroid stimulating hormone increased (Investigations) | 4 (4) | 2 (2)
Blood urea increased (Investigations) | 5 (5) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 2 (2)
Lymphocyte count decreased (Investigations) | 7 (9) | 1 (1)
Neutrophil count decreased (Investigations) | 6 (10) | 5 (15)
Thyroxine free increased (Investigations) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 18 (22) | 4 (5)
Weight increased (Investigations) | 3 (4) | 2 (2)
White blood cell count decreased (Investigations) | 13 (26) | 4 (15)
Decreased appetite (Metabolism and nutrition disorders) | 15 (20) | 8 (12)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (9)
Hyperuricaemia (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 25 (33) | 4 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 12 (15) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 20 (40) | 8 (10)
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 (18) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (8) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (15) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 9 (10) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (3)
Haematuria (Renal and urinary disorders) | 4 (4) | 3 (4)
Proteinuria (Renal and urinary disorders) | 6 (6) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 8 (9) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (18) | 5 (7)
Rash (Skin and subcutaneous tissue disorders) | 18 (18) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2)
Hypertension (Vascular disorders) | 5 (7) | 2 (2)
Lymphoedema (Vascular disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights

DOCUMENTS (2):
  • Study Protocol (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT04693234/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT04693234/SAP_001.pdf